CLINICAL TRIAL: NCT01069016
Title: Comparison of Sacral Nerve Modulation and Pudendal Nerve Stimulation in Treatment of Fecal Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Principal Investigator, Lukas Marti, Leitender Arzt, Cantonal Hospital of St. Gallen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SNS/PNS
Record Dates: First submitted 2010-02-11; First posted 2010-02-17 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Fecal Incontinence
Keywords: Fecal Incontinence; Colorectal surgery; Sacral nerve stimulation; Pudendal nerve stimulation
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sacral nerve modulation first (Experimental): Sacral nerve modulation is applied before the pudendal nerve stimulation. There is no "wash-out" period (pause) between the two treatments.
  Interventions: Procedure: Sacral nerve modulation; Procedure: Pudendal nerve stimulation
- Pudendal nerve stimulation first (Experimental): Pudendal nerve stimulation is applied before the sacral nerve modulation. There is no "wash-out" period (pause) between the two treatments.
  Interventions: Procedure: Sacral nerve modulation; Procedure: Pudendal nerve stimulation

INTERVENTIONS:
Procedure: Sacral nerve modulation — For one week the sacral nerve is continuously stimulated by an external pulse generator. Strength of stimulation can be adjusted by the patient.
  Other Names: SNM; Sacral nerve stimulation; SNS
Procedure: Pudendal nerve stimulation — For one week the pudendal nerve is continuously stimulated by an external pulse generator. Strength of stimulation can be adjusted by the patient.
  Other Names: PNS

SUMMARY:
Sacral nerve modulation (SNM) is an established treatment for refractory lower urinary tract and bowel dysfunction (Spinelli 2008). Pudendal nerve stimulation (PNS) has been proposed for patients failing SNM treatment of urinary dysfunction (Spinelli 2005). In this study SNM and PNS are compared for the treatment of fecal incontinence. In a test phase, both treatments will be applied for one week each in a randomized and blinded order (cross-over design). After the test phase the more successful treatment will be determined and applied permanently. If both treatments are equally sufficient, PNS will be chosen for permanent stimulation, since preliminary data indicate that PNS has a lower power consumption than SNM. Lower power consumption results in a longer lifetime of the stimulator, thus requiring less replacement surgeries.

DETAILED DESCRIPTION:
Primary Surgery:

* Implantation of two electrodes, one placed next to the sacral nerve, one close to the pudendal nerve. Electrode wires are passed through the skin just above the gluteal region and are marked S and P. One of the sub-investigators (not involved in the follow-up) replaces the S and P marks by 1 and 2 marks in absence of the operating surgeon. Assignment of 1 and 2 is carried out in a predefined randomized fashion (computerized block randomization).

Test phase:

* Electrode labeled 1 is connected to a stimulator and the nerve is stimulated for one week, then the other electrode is stimulated for a week.
* Based on bowel habit diary, Wexner score (Jorge 1993) and subjective experience of the patient, the more successful treatment is chosen. If both electrodes were equally successful, the pudendal nerve electrode will be chosen for permanent stimulation.

Secondary surgery:

* After unblinding, the less effective electrode is removed and the remaining electrode is connected to an implanted stimulator (permanent phase). In case both treatments were unsuccessful, both electrodes are removed.

ELIGIBILITY:
Inclusion Criteria:

* fecal incontinence nonresponsive to conservative treatment

Exclusion Criteria:

* sacral or perineal infection
* sphincter defect larger than 60° (sonography)
* pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-02 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Power consumption of stimulator | 14 days

SECONDARY OUTCOMES:
Wexner Score (Jorge 1993) | 7, 14 days, 3, 6 & 12 months
Incidence of surgical complications (adverse events) graded according to Dindo (2004) | 30 days
Quality of Life (FIQL (Rockwood 2000)) | 14 days, 3, 6 & 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Lukas Marti, MD, Principal Investigator — Dep. of Surgery, Cantonal Hospital St. Gallen
Locations (1):
- Department of Surgey, Cantonal Hospital St. Gallen, Sankt Gallen, Switzerland

REFERENCES:
- [Background] Spinelli M, Sievert KD. Latest technologic and surgical developments in using InterStim Therapy for sacral neuromodulation: impact on treatment success and safety. Eur Urol. 2008 Dec;54(6):1287-96. doi: 10.1016/j.eururo.2008.01.076. Epub 2008 Feb 8. PMID 18336992
- [Background] Spinelli M, Malaguti S, Giardiello G, Lazzeri M, Tarantola J, Van Den Hombergh U. A new minimally invasive procedure for pudendal nerve stimulation to treat neurogenic bladder: description of the method and preliminary data. Neurourol Urodyn. 2005;24(4):305-9. doi: 10.1002/nau.20118. PMID 15977260
- [Background] Jorge JM, Wexner SD. Etiology and management of fecal incontinence. Dis Colon Rectum. 1993 Jan;36(1):77-97. doi: 10.1007/BF02050307. PMID 8416784
- [Background] Rockwood TH, Church JM, Fleshman JW, Kane RL, Mavrantonis C, Thorson AG, Wexner SD, Bliss D, Lowry AC. Fecal Incontinence Quality of Life Scale: quality of life instrument for patients with fecal incontinence. Dis Colon Rectum. 2000 Jan;43(1):9-16; discussion 16-7. doi: 10.1007/BF02237236. PMID 10813117
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- See also: Proctological consultations, Department of Surgery — http://www.chirurgie.kssg.ch/home/unsere_klinik/Leistungsangebot_standort_st_gallen/koloproktologie.html